CLINICAL TRIAL: NCT03237026
Title: Decipher the Biology of Lethal Prostate Cancer-Using Urine Metabolomics and Proteomics Profiling to Search for Predictive and Prognostic Markers for Treatment Outcomes in Prostate Cancer Patients
Brief Title: Predictive and Prognostic Markers for Treatment Outcomes in Prostate Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201705032RINA
Record Dates: First submitted 2017-07-30; First posted 2017-08-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostatectomy; prostate radiotherapy; chemotherapy; immunotherapy; biomarkers; metabolomics; proteomics; urine
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: fresh urine samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: Ttaining chort will be recruited in the first 36 months of the study period to generate the first batch of urine metabolomic and proteomic profiles as predictive and prognostic markers.
  Interventions: Other: No intervention required
- Cohort B: Validation cohort will be recruited in the next 24 months of the study period .
  Interventions: Other: No intervention required

INTERVENTIONS:
Other: No intervention required — No intervention required

SUMMARY:
The study aims to identify potential urine marker metabolites as predictive or prognostic markers for treatment outcomes in patients with prostate cancer.

DETAILED DESCRIPTION:
This is a single-center single-arm translational study where patients with prostate cancer who are about to receive definitive treatments will be invited to participate the study. After signing the approved informed consent, eligible and consenting subjects will donate their fresh urine samples for subsequent untargeted metabolomics and proteomics study to identify potential metabolite and protein markers that are able to predict responses (including efficacy and side effects) to definitive treatments. All subjects who have received varied treatment before the study can NOT be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have histopathologically confirmed prostate adenocarcinoma.
2. Subjects who age 30 years to 100 years
3. Subjects who agree to undergo the any of the following four treatments, including radical prostatectomy, definitive prostate radiotherapy, systemic chemotherapy, and androgen deprivation therapy for prostate cancer.
4. Subjects who understand and will comply with the entire study procedures, consent to donate his spot urine (once for 50 ml) for urine metabolomics and proteomic profiling, and agree with subsequent collection and analysis of his clinical information including results of biopsy and the details of treatments and outcomes. (Note: Subjects will be told that the urine metabolomics and proteomics results will not be revealed to them.)

Exclusion Criteria:

1. Subjects who have other cancers that have not been curatively treated or are disease-free for only 3 years or less. Subjects who have other genitourinary cancers (urothelial, renal cell, etc) are NOT allowed no matter what the disease-free duration is. However, subjects who have been curatively treated and are disease-free for 3 years or longer are allowed to be enrolled.
2. Subjects who have severe organ function impairment which may significantly alter general cell metabolism or proteomics profiles determined by the investigators, such as Cre > 3.0, HbA1c > 9.0%, symptomatic heart failure, or other symptomatic metabolic diseases.
3. Subjects who have significant infection or inflammation within 8 weeks of the biopsy.
4. Subjects who are taking medicine(s) that may, deemed by the investigators, substantially affect cell metabolism and proteomics profiles.
5. Subjects who have a life expectancy less than 12 months.

Ages: 30 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A. Expected subject number to be enrolled: 360 men at NTUH.
  1. Radical prostatectomy (OP, N=100): 50 subjects each for Cohort A and Cohort B, respectively.
  2. Radiotherapy (RT, N=140): 70 subjects each for Cohort A and Cohort B, respectively.
  3. Androgen-deprivation therapy (ADT, N=60): 30 subjects each for Cohort A and Cohort B, respectively
  4. Systemic chemotherapy (Chemo, N=60): 30 subjects for Cohort A and Cohort B, respectively
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2017-10-11 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
Biochemical recurrence or progression | 5 years
toxicity profile, survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yeong-Shiau Pu, MD PhD, Principal Investigator — Department of Urology, National Taiwan University Hospital
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No